CLINICAL TRIAL: NCT00047112
Title: Randomized Study of Pre-Operative Radio-Chemotherapy Versus Surgery Alone in Thoracic Esophageal Cancer Deemed to be Resectable
Brief Title: Surgery With or Without Radiation Therapy and Chemotherapy in Treating Patients With Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Collaborators: GERCOR - Multidisciplinary Oncology Cooperative Group (Other); European Organisation for Research and Treatment of Cancer - EORTC (Network); UNICANCER (Other); Societe Francaise de Radiotherapie Oncologique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000257600; FFCD-9901; EORTC-22001; EORTC-40001; FRE-FNCLCC-FFCD-9901; FRE-GERCOR-FFCD-9901; SFRO-FFCD-9901; EU-20215
Record Dates: First submitted 2002-10-03; First posted 2003-01-27 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Esophageal Cancer
Keywords: adenocarcinoma of the esophagus; squamous cell carcinoma of the esophagus; stage I esophageal cancer; stage II esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Cisplatin; Fluorouracil; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHIMIORADIOTHERAPIE SUIVIE DE CHIRURGIE (Experimental): CHIMIORADIOTHERAPIE SUIVIE DE CHIRURGIE
  Interventions: Drug: cisplatin; Drug: fluorouracil; Procedure: conventional surgery; Procedure: neoadjuvant therapy; Radiation: radiation therapy
- CHIRURGIE SEULE (Active Comparator): CHIRURGIE SEULE
  Interventions: Procedure: conventional surgery

INTERVENTIONS:
Drug: cisplatin
  Arms: CHIMIORADIOTHERAPIE SUIVIE DE CHIRURGIE
Drug: fluorouracil
  Arms: CHIMIORADIOTHERAPIE SUIVIE DE CHIRURGIE
Procedure: conventional surgery
Procedure: neoadjuvant therapy
  Arms: CHIMIORADIOTHERAPIE SUIVIE DE CHIRURGIE
Radiation: radiation therapy
  Arms: CHIMIORADIOTHERAPIE SUIVIE DE CHIRURGIE

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving combination chemotherapy with radiation therapy before surgery may shrink the tumor so it can be removed during surgery. It is not yet known if surgery is more effective with or without radiation therapy and chemotherapy in treating esophageal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery with or without radiation therapy and chemotherapy in treating patients who have esophageal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with resectable thoracic esophageal cancer treated with neoadjuvant radio-chemotherapy and surgery versus surgery alone.
* Compare the disease-free survival of patients treated with these regimens.
* Compare the surgical mortality and morbidity of patients treated with these regimens.
* Compare the resectability of patients treated with these regimens.
* Determine the validation of new prognostic factors for survival of these patients and/or the efficacy of this neoadjuvant treatment.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to histology (epidermoid carcinoma vs adenocarcinoma vs undifferentiated carcinoma), stage (I vs IIA vs IIB), tumor location (above the carina vs below the carina), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy daily 5 days a week for 5 weeks. Patients receive fluorouracil IV continuously on days 1-4 and 29-32 and cisplatin IV on days 1 or 2 and 29 or 30 (or a lower dose on days 1-5 and 29-33). Within 4-8 weeks after completion of radio-chemotherapy, patients undergo surgical resection.
* Arm II: Patients undergo surgical resection. Patients are followed every 4 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 380 patients (190 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage I or II thoracic esophageal cancer

  * Tumor no greater than 3 cm with no invasion of mediastinal structures with or without extension to the lymph nodes (T1-2, N0-1, M0) OR
  * Tumor greater than 3 cm with no invasion of mediastinal structures and no adenopathy greater than 1 cm (T3, N0, M0)
  * Epidermoid carcinoma or adenocarcinoma
* Previously untreated
* Deemed resectable with curative intent
* No carcinoma in situ
* No small cell anaplastic carcinoma (i.e., chromogranin negative)
* No small cell neuroendocrine carcinoma (i.e., chromogranin positive)
* No multifocal esophageal carcinoma (i.e., 2 or more distinct lesions 5 or more cm apart)
* No involvement of the pharyngoesophageal junction and the first 4 cm of the esophagus (i.e., where the proximal edge of the tumor is less than 19 cm from the dental arch)
* No evidence of extension to the tracheobronchial tree at endoscopy, ultrasound, or CT scan (simple compression allowed)
* No signs of mediastinal involvement on CT scan
* No palpable subclavicular lymph nodes or involvement after cytology needle aspiration
* No lymph nodes from the origin of the celiac greater than 1 cm on CT scan

  * Perigastric lymph nodes far from the celiac trunk and deemed resectable allowed unless tumor is more than 30 mm on CT scan

PATIENT CHARACTERISTICS:

Age

* Under 75

Performance status

* WHO 0-1

Life expectancy

* Not specified

Hematopoietic

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* SGOT/SGPT ratio no greater than 1
* Albumin at least 35 g/L
* Total protein greater than 80%
* No liver cirrhosis with previous failure
* No ascites
* No jaundice
* No rupture of varicose esophageal veins
* No presence of varicose esophageal veins

Renal

* Creatinine no greater than 1.25 times normal

Cardiovascular

* Arterial O_2 greater than 60 mm Hg
* Arterial CO_2 no greater than 45 mm Hg
* No myocardial infarction within the past 6 months
* No progressive coronary artery disease grade 2 or greater
* No recent left ventricular failure
* No arterial disease stage II-IV

Pulmonary

* FEV_1 greater than 1 L/sec

Other

* Able to receive either study treatment
* No recurrent paralysis
* No weight loss greater than 10% from baseline
* No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* Not pregnant
* Fertile patients must use effective contraception during and for 3 months after completion of chemotherapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2002-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
overal survival | 2010

SECONDARY OUTCOMES:
recurrence free survival | 2010

CONTACTS AND LOCATIONS:
Overall Officials: J. P. Triboulet, Study Chair — Centre Hospitalier Regional et Universitaire de Lille; Jean-Francois Seitz, MD, Study Chair — Institut Paoli-Calmettes
Locations (73):
- Belgium (5):
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universiteit Gent, Ghent
  - CHR - Clinique Saint Joseph - Hopital de Warqueguies, Mons
- France (63):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Centre Paul Papin, Angers
  - Arras
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - CHU Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Docteur Duchenne, Boulogne-sur-Mer
  - C.H. Bourg En Bresse, Bourg-en-Bresse
  - Centre Hospitalier de Bourgoin - Jallieu, Bourgoin
  - CHU Brest - Hopital De La Cavale Blanche, Brest
  - Centre Hospitalier General, Brivé
  - CHU de Caen, Caen
  - Clinique Sainte Marie, Chalon-sur-Saône
  - CHR Clermont Ferrand, Hotel dieu, Clermont-Ferrand
  - Hopital Beaujon, Clichy
  - Hopital Louis Pasteur, Colmar
  - Centre Hospitalier de Lagny, Compiègne
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre Hospitalier De Dunkerque - CHD, Dunkirk
  - Évreux
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Hopital Andre Mignot, Le Chesnay
  - Centre Jean Bernard, Le Mans
  - Hopital Robert Boulin, Libourne
  - Polyclinique Du Bois, Lille
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Hopital de la Croix Rousse, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Assistance Publique Hopitaux de Marseille Hopitaux Sud, Marseille
  - CHU de la Timone, Marseille
  - Centre Gray, Maubeuge
  - Centre Hospitalier de Meaux, Meaux
  - Hopital Notre-Dame de Bon Secours, Metz
  - CH Meulan, Meulan-en-Yvelines
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Hospitalier, Mulhouse
  - CHR Hotel Dieu, Nantes
  - Hopital de l'Archet, Nice
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Saint Antoine, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital Jean Bernard, Poitiers
  - Centre Hospitalier De Pontivy, Pontivy
  - Institut Jean Godinot, Reims
  - Centre Hospitalier Universitaire, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier D'Agen, Saint-Esprit
  - Centre Hospitalier Intercommunal de Poissy, Saint-Germain-en-Laye
  - Centre Joliot Curie Des Docteurs Jean-Christophe Chardon Jacques Hernandez Et Laurent Gasnault, Saint-Martin-Boulogne
  - Clinique Sainte Clotilde, Sainte-Clotilde
  - C.H. Senlis, Senlis
  - Centre Hospitalier General De Saint-Malo, St-Malo
  - Centre Paul Strauss, Strasbourg
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Hopital Universitaire Hautepierre, Strasbourg
  - CHU de Tours, Tours
  - Nouvelle Clinique Generale, Valence
  - Centre Hospitalier de Valenciennes, Valenciennes
  - CHU de Nancy - Hopitaux de Brabois, Vandœuvre-lès-Nancy
  - Centre d'Oncologie Saint-Yves, Vannes
  - Institut Gustave Roussy, Villejuif
- Germany (4):
  - Robert Roessle Comprehensive Cancer Center at University of Berlin - Charite Campus Buch, Berlin
  - Universitaet Erlangen, Erlangen
  - Klinikum der Albert - Ludwigs - Universitaet Freiburg, Freiburg im Breisgau
  - Universitaets-Krankenhaus Eppendorf, Hamburg
- Academisch Ziekenhuis Maastricht, Maastricht, Netherlands

REFERENCES:
- [Background] Mariette C, Robb WB, Piessen G. Reply to Letter: "The Role of Surgery for Patients With a Complete Clinical Response After Chemoradiation for Esophageal Cancer". Ann Surg. 2015 Dec;262(6):e101-2. doi: 10.1097/SLA.0000000000000668. No abstract available. PMID 24670853
- [Result] Mariette C, Dahan L, Mornex F, Maillard E, Thomas PA, Meunier B, Boige V, Pezet D, Robb WB, Le Brun-Ly V, Bosset JF, Mabrut JY, Triboulet JP, Bedenne L, Seitz JF. Surgery alone versus chemoradiotherapy followed by surgery for stage I and II esophageal cancer: final analysis of randomized controlled phase III trial FFCD 9901. J Clin Oncol. 2014 Aug 10;32(23):2416-22. doi: 10.1200/JCO.2013.53.6532. Epub 2014 Jun 30. PMID 24982463
- [Result] Robb WB, Dahan L, Mornex F, Maillard E, Thomas PA, Meunier B, Boige V, Pezet D, Le Brun-Ly V, Bosset JF, Mabrut JY, Triboulet JP, Bedenne L, Seitz JF, Mariette C; Federation Francaise de Cancerologie Digestive, Societe Francaise de Radiotherapie Oncologique, Union des Centres de Lutte Contre le Cancer, Groupe Cooperateur Multidisciplinaire en Oncologie, French EsoGAstric Tumour working group, Federation de Recherche En Chirurgie. Impact of neoadjuvant chemoradiation on lymph node status in esophageal cancer: post hoc analysis of a randomized controlled trial. Ann Surg. 2015 May;261(5):902-8. doi: 10.1097/SLA.0000000000000991. PMID 25361220
- [Derived] Robb WB, Messager M, Dahan L, Mornex F, Maillard E, D'Journo XB, Triboulet JP, Bedenne L, Seitz JF, Mariette C; Federation Francophone de Cancerologie Digestive; Societe Francaise de Radiotherapie Oncologique; Union des Centres de Lutte Contre le Cancer; Groupe Cooperateur Multidisciplinaire en Oncologie; French EsoGAstric Tumour working group - Federation de Recherche En Chirurgie. Patterns of recurrence in early-stage oesophageal cancer after chemoradiotherapy and surgery compared with surgery alone. Br J Surg. 2016 Jan;103(1):117-25. doi: 10.1002/bjs.9959. Epub 2015 Oct 29. PMID 26511668